CLINICAL TRIAL: NCT04013490
Title: Safety Evaluation and Effect of Food Supplement Containing Dietary Fiber From Cassava on the Alterations of Physiological Parameters in Overweight Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Jintanaporn Wattanathorn, Associated Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HE611054
Record Dates: First submitted 2019-06-20; First posted 2019-07-09 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Overweight
Keywords: physiological parameters; consumption safety; cassava; food supplement; overweight female
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo capsule (Placebo Comparator): Subject receive the Placebo product for 4 weeks.
  Interventions: Dietary Supplement: Cassava dietary fiber capsule
- Cassava dietary fiber capsule 1.5 g/day (Active Comparator): Subjects receive Cassava dietary fiber capsule at the dose of 1.5 g/day for 4 weeks.
  Interventions: Dietary Supplement: Cassava dietary fiber capsule
- Cassava dietary fiber capsule 3 g/day (Active Comparator): Subjects receive Cassava dietary fiber capsule at the dose of 3 g/day for 4 weeks.
  Interventions: Dietary Supplement: Cassava dietary fiber capsule

INTERVENTIONS:
Dietary Supplement: Cassava dietary fiber capsule — Cassava dietary fiber capsule or placebo will be consumed once daily at the recommended doses of each group.

SUMMARY:
This study is set up to determine the consumption safety and the effect of a food supplement containing dietary fiber from cassava on the alterations of physiological parameters including fasting blood sugar, HbA1c, insulin resistance, lipid profiles, atherogenic index, blood pressure and gut microbes in overweight female volunteers.

DETAILED DESCRIPTION:
Cassava is one of the important industrial crops in Thailand. The leftover fiber of cassava is still valuable and can be used as a dietary fiber. The previous study demonstrated that dietary fiber containing cassava fiber was safe for consumption without any contamination of the cyanide and heavy metals. Moreover, the microbial contaminations were within the safety range. The toxicity study revealed that the LD50 of the cassava dietary fiber was more than 5 g/kg body weight (BW) and NOAEL was 3 g/kg BW. The NOAEL was used to calculate the human equivalent dose for determining the effect of cassava dietary fiber in a clinical study.

Cassava dietary fiber consists of water-insoluble fiber such as cellulose more than 50%. The previous study showed that insoluble fiber decreased the risk of type 2 diabetes and increased insulin release. Moreover, a high fiber diet also decreased the fasting glucose and HbA1C in type 2 diabetes volunteer. In addition, the effect of dietary fiber on the reduction of cholesterol was also reported. The previous study reported that the cassava dietary fiber could decrease the total cholesterol, triglyceride but increase high-density lipoprotein in a dyslipidemia rat model. Therefore, the cassava fiber might be the potential food supplement for the control of blood sugar and lipid profiles in human. However, less scientific data support the effect of cassava dietary fiber in human.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women age between 35-60 years old
* BMI 23-29.99
* Blood pressure <140/90 mmHg
* Fasting plasma glucose < 100 mg/dL

Exclusion Criteria:

* Presence of any chronic diseases
* Alcohol addict or consume more than 2 units/day
* Smoking more than 10 cigarettes per day
* Medication or herbal medicine usage within 1 month prior to the study
* Use any medication or food supplement which affect to outcomes
* Pregnant or breastfeeding women
* Athlete

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
The fasting blood sugar level | Baseline and 4 weeks of intervention
  The previous study reported that high dietary fiber could decrease the fasting blood sugar in type 2 diabetes patient. The overweight female volunteer receive food supplement containing dietary fiber from Cassava should show the lower level of fasting blood sugar than the placebo-treated group after 4 weeks of intervention.
The atherogenic index | 4 weeks of intervention
  The atherogenic index is an index composed of triglycerides and high-density lipoprotein cholesterol. It has been used to quantify blood lipid levels and commonly used as an optimal indicator of dyslipidemia and associated diseases. The food supplement containing dietary fiber from Cassava might be able to decrease the atherogenic index in overweight female volunteer. The overweight female volunteer receive food supplement containing dietary fiber from Cassava should show the lower number of the atherogenic index than the placebo-treated group after 4 weeks of intervention.

SECONDARY OUTCOMES:
hemoglobin A1c concentration | 4 weeks of intervention
  A hemoglobin A1c (HbA1c) test measures the amount of blood sugar (glucose) attached to hemoglobin. This result shows the average amount of glucose attached to hemoglobin has been over the past three months. The previous study reported that high dietary fiber could decrease the HbA1C in type 2 diabetes patient. The food supplement containing dietary fiber from Cassava might be able to decrease the HbA1C in overweight female volunteer. The overweight female volunteer receive food supplement containing dietary fiber from Cassava should show the lower HbA1C level than the placebo-treated group after 4 weeks of intervention.
Homeostasis model assessment-insulin resistance (HOMA-IR) | 4 weeks of intervention
  HOMA-IR was computed with the formula: fasting plasma glucose (mmol/l) multiplied fasting serum insulin (mU/l) divided by 22.5. Low HOMA-IR values indicate high insulin sensitivity, whereas high HOMA-IR values indicate low insulin sensitivity (insulin resistance). The overweight female volunteers receive food supplement containing dietary fiber from Cassava should show the lower HOMA-IR than the placebo-treated group after 4 weeks of intervention.
Low-density lipoprotein (LDL) concentration | 4 weeks of intervention
  LDL is considered bad cholesterol and a leading cause of atherosclerosis formation. The food supplement containing dietary fiber from Cassava might be able to decrease the LDL level in overweight female volunteer. The overweight female volunteers receive food supplement containing dietary fiber from Cassava should show the lower LDL concentration than the placebo-treated group after 4 weeks of intervention.
High-density lipoprotein (HDL) concentration | 4 weeks of intervention
  HDL is considered as good cholesterol and believed that it acts as a scavenger and carrying of LDL from the arteries back to the liver. The food supplement containing dietary fiber from Cassava might be able to increase the LDL level in overweight female volunteer. The overweight female volunteers receive food supplement containing dietary fiber from Cassava should show a higher HDL concentration than the placebo-treated group after 4 weeks of intervention.
Triglyceride (TG) concentration | 4 weeks of intervention
  TG is one type of fat in the blood which converted from the excess energy from the diet. A high triglyceride level combined with high LDL (bad) cholesterol or low HDL (good) cholesterol is linked with fatty buildups within the artery walls, which increases the risk of heart attack and stroke in an overweight person. The food supplement containing dietary fiber from Cassava might be able to decrease the LDL level in overweight female volunteer. The overweight female volunteers receive food supplement containing dietary fiber from Cassava should show the lower TG concentration than the placebo-treated group after 4 weeks of intervention.
Cholesterol concentration | 4 weeks of intervention
  The high level of cholesterol is a cause of atherosclerosis in the blood vessel. The food supplement containing dietary fiber from Cassava might be able to decrease the cholesterol level in overweight female volunteer. The overweight female volunteers receive food supplement containing dietary fiber from Cassava should show the lower cholesterol concentration than the placebo-treated group after 4 weeks of intervention.
Body mass index (BMI) | 4 weeks of intervention
  The food supplement containing dietary fiber from Cassava might be able to decrease the BMI in overweight female volunteer. The overweight female volunteers receive food supplement containing dietary fiber from Cassava should show the lower BMI than the placebo-treated group after 4 weeks of intervention.
Gut microbes | 4 weeks of intervention
  It has been reported that the dysbiosis can cause the alteration of glucose metabolism, lipid metabolism, and dyslipidemia. Moreover, the high fiber diet causes the elevation of good bacteria in the gut and exert many effects. The food supplement containing dietary fiber from Cassava might be able to increase the good gut microbes in overweight female volunteer. The overweight female volunteers receive food supplement containing dietary fiber from Cassava should show higher gut microbes than the placebo-treated group after 4 weeks of intervention.
The consumption safety of food supplement containing dietary fiber from Cassava using Systolic and Diastolic Blood pressure | 4 weeks of intervention
  If the supplement containing dietary fiber from Cassava is safe, the blood pressure should be within the normal range.
The consumption safety of food supplement containing dietary fiber from Cassava using the electrocardiogram pattern and QT interval data | 4 weeks of intervention
  If the supplement containing dietary fiber from Cassava is safe, the EKG pattern and the QT interval should be within the normal range.
Consumption safety of food supplement containing dietary fiber from Cassava using blood chemistry | 4 weeks of intervention
  The blood chemistry values including renal function test, liver function test, and electrolytes will be determined and the data will be expressed as the number of subjects presented with abnormal blood chemistry value.
Consumption safety of food supplement containing dietary fiber from Cassava using hematolgical values. | 4 weeks of intervention
  The hematological values including red blood cell, white blood cell, hematocrit, and platelet will be determined and the data will be expressed as a number of subjects presented with abnormal hematological value.

CONTACTS AND LOCATIONS:
Locations (1):
- Jitanaporn Wattanathorn, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No